CLINICAL TRIAL: NCT02522715
Title: A Phase I/II Trial of Concurrent Chemohormonal Therapy Using Enzalutamide (MDV-3100) and Cabazitaxel in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Enzalutamide and Cabazitaxel in Treating Patients With Metastatic, Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Julie Graff, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00011227; NCI-2015-01103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11227; CRS00001390; IRB00011227 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2015-07-24; First posted 2015-08-13 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; enzalutamide; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabazitaxel, enzalutamide) (Experimental): Patients receive cabazitaxel IV over 1 hour on day 1 and enzalutamide PO QD on days 1-21 (days 2-21 of cycle 1). Patients also receive prednisone PO BID as standard of care with cabazitaxel. Cycles repeat every 21 days for 6-10 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue enzalutamide PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabazitaxel; Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Prednisone

INTERVENTIONS:
Drug: Cabazitaxel — Given IV
  Other Names: Jevtana; RPR-116258A; Taxoid XRP6258; XRP-6258
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone

SUMMARY:
This phase I/II trial studies the side effects and best dose of cabazitaxel when given together with enzalutamide in treating patients with prostate cancer that has spread to other places in the body (metastatic) and has not responded to treatment with hormones or no longer responds to treatment with hormones (hormone-resistant). Drugs used in chemotherapy, such as cabazitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Androgen can cause the growth of prostate cancer cells. Hormone therapy using enzalutamide may fight prostate cancer by blocking the use of androgen by the tumor cells. Giving cabazitaxel together with enzalutamide may work better in treating metastatic, hormone-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of combination treatment with enzalutamide and cabazitaxel (as determined by percent dose limiting toxicities [DLT], where DLT < 17% is consistent with it being a tolerable combination).

II. To determine the efficacy of treatment with the hormonal agent enzalutamide and the chemotherapy cabazitaxel in combination in men with metastatic castration-resistant prostate cancer (CRPC) (as determined by percent of patients achieving >= 90% prostate specific antigen [PSA] declines following initiation of treatment).

SECONDARY OBJECTIVES:

I. To further define the anticancer effect and safety profile of the combination of enzalutamide and cabazitaxel.

Ia. Collect toxicity data (description of adverse events). Ib. Determine PSA response (percent of patients who achieve >= 50% PSA decline and >= 30% PSA decline).

Ic. Examine pharmacokinetic (PK) data of cabazitaxel to characterize enzalutamide and cabazitaxel pharmacokinetic blood levels.

Id. Determine tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for measurable disease and Prostate Cancer Working Group 2 criteria for non-measurable (bone) disease.

Ie. Determine overall survival.

EXPLORATORY OBJECTIVES:

I. To determine baseline (and at progression) biological tumor characteristics to evaluate for possible biomarkers indicative or predictive of response: apoptosis by cleaved caspase 3; androgen signaling axis (including but not limited to: androgen receptor expression, androgen receptor splice variants, and intratumoral androgen levels), and glucocorticoid receptor.

II. To collect circulating tumor cells (CTCs) and determine the degree to which tumor characteristics (delineated above) are shared by the CTCs.

III. To collect plasma and serum pre-treatment and at progression for assessment of circulating micro-ribonucleic acid (RNA)s and other circulating markers.

IV. To collect buffy coat to evaluate for steroid transporters.

OUTLINE: This is a dose de-escalation study of cabazitaxel.

Patients receive cabazitaxel intravenously (IV) over 1 hour on day 1 and enzalutamide orally (PO) once daily (QD) on days 1-21 (days 2-21 of cycle 1). Patients also receive prednisone PO twice daily (BID) as standard of care with cabazitaxel. Cycles repeat every 21 days for 6-10 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue enzalutamide PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic CRPC
* Willing to provide a tumor sample via biopsy from a metastatic site of disease to be collected at screening if safe and feasible per discretion of treating investigator; adequate archival metastatic tissue can be used, if available, in lieu of baseline biopsy if done when patient had CRPC; patients without a site amenable to biopsy and lack of archival tissue may still join the study
* Evidence of prostate cancer progression by any of the following criteria: radiographic or PSA criteria, or symptomatic progression related to prostate cancer
* Castrate testosterone levels (< 50 ng/dL) achieved by orchiectomy or maintenance on a luteinizing hormone-releasing hormone (LHRH) agonist or antagonist
* Histologic confirmation of original prostate cancer diagnosis per institutional standard; life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin within normal institutional limits (or < 2 X the upper limit of normal in those with Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 X institutional upper limit of normal
* Creatinine within less than the institutional upper limit of normal
* Creatinine clearance >= 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Subject agrees to use a double barrier method of birth control during the course of study treatment period with enzalutamide and/or cabazitaxel treatment and for at least 3 months after the study is discontinued

  * A double-barrier method of contraception involves the use of a condom in combination with 1 of the following: contraceptive sponge, diaphragm, or cervical ring with spermicidal gel or foam
  * Subject who has had a vasectomy at least 6 months prior to starting study treatment period and those whose female sexual partner(s) are more than 55 years of age and postmenopausal for at least 2 years or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) agree to use at least a condom
* Ability to understand, and the willingness to sign, a written informed consent document, as well as comply with study requirements
* Must have appropriate wash out (> 6 half-lives) of androgen receptor antagonists, 5 alpha reductase inhibitors or ketoconazole prior to the start of cycle 1; if the agent is not in the table below, the washout should be 2 weeks

  * Bicalutamide; approximate half-life: 6 days; washout period required: 36 days
  * Flutamide; approximate half-life: 6 hours; washout period required: 36 hours
  * Nilutamide approximate half-life: 4 days; washout period required: 24 days
  * Finasteride; approximate half-life: 8 hours; washout period required: 48 hours
  * Aminoglutethimide; approximate half-life: 15 hours; washout period required: 4 days
  * Ketoconazole; approximate half-life: 8 hours; washout period required: 48 hours

Exclusion Criteria:

* Prior chemotherapy for mCRPC prostate cancer; chemotherapy given neoadjuvantly, adjuvantly, or for hormone sensitive metastatic disease is permitted as long as the cancer did not progress on chemotherapy AND > 6 months have elapsed
* Patients may not have received any other investigational agents within the last 14 days at the time of treatment start
* Patients may not have received enzalutamide or ARN-509 (another androgen receptor antagonist) in the past
* Patients may not have received cabazitaxel in the past
* Subject has clinical signs suggestive of high or imminent risks for pathological fracture, spinal cord compression and/or cauda equina syndrome
* History of severe hypersensitivity reaction (>= grade 3) to docetaxel, polysorbate 80 containing drugs, or any of the capsule components of enzalutamide, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 family 3, subfamily A, polypeptide 4/5 (3A4/5); (a one-week wash-out period is necessary for patients who are already on these treatments)
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled diabetes, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subject has a history of seizure or any condition that may predispose to seizure including, but not limited to, underlying brain injury, stroke in the past 6 months, primary brain tumors, brain metastases, prior seizures
* Subject has a history of unexplained loss of consciousness or transient ischemic attack within 12 months of treatment start
* Subject is unwilling to stop using herbal supplements that can affect the PSA, such as saw palmetto or prostate cancer (PC)-SPES
* Subject has another active malignancy other than non-melanomatous skin cancer (unless it is metastatic) or superficial bladder cancer
* Must not have a gastrointestinal condition that would interfere with absorption
* Subjects may not be on other therapies that affect hormone levels, such as estrogens, testosterones, ketoconazole during this study; however, megestrol for hot flashes is permitted

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2026-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Julie N Graff, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I accrual occurred between November 2015 and April 2016. Phase II accrual occurred between January 2017 and March 2019. The last follow-up date is anticipated to be December 2023.
Pre-assignment Details: One participant withdrew before receiving study treatment and was therefore excluded from safety and efficacy analysis.
Groups:
- Phase I - Treatment (Cabazitaxel, Enzalutamide); Phase II - Treatment (Cabazitaxel, Enzalutamide): Patients receive 25 mg/m2 cabazitaxel IV over 1 hour on day 1 and enzalutamide PO QD on days 1-21 (days 2-21 of cycle 1). Patients also receive prednisone PO BID as standard of care with cabazitaxel. Cycles repeat every 21 days for 6-10 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue enzalutamide PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
  Cabazitaxel: Given IV
  Enzalutamide: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Prednisone: Given PO
Period: Overall Study
Arm/Group | Phase I - Treatment (Cabazitaxel, Enzalutamide) | Phase II - Treatment (Cabazitaxel, Enzalutamide)
Started | 3 | 33 (+1 early withdrawal)
Completed | 3 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II - Treatment (Cabazitaxel, Enzalutamide): Patients receive 25 mg/m2 cabazitaxel IV over 1 hour on day 1 and enzalutamide PO QD on days 1-21 (days 2-21 of cycle 1). Patients also receive prednisone PO BID as standard of care with cabazitaxel. Cycles repeat every 21 days for 6-10 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue enzalutamide PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase I - Treatment (Cabazitaxel, Enzalutamide) | Phase II - Treatment (Cabazitaxel, Enzalutamide) | Total
Number analyzed (Participants) | 3 | 33 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 7 | 8
  >=65 years | 2 | 26 | 28
Age, Continuous [Median (Full Range); unit: years] | 66 [47 to 78] | 69 [51 to 82] | 69 [47 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 33 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 3 | 28 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 33 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting ToxicitiesGgraded by National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (Phase I)
Description: The percentage of participants will be reported with 95% confidence interval using exact method.
Time Frame: Up to 42 days
Population: Patients with metastatic CRPC. Phase I patients who received at least two cycles of study drugs will be evaluable for DLT analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I - Treatment (Cabazitaxel, Enzalutamide)
Number analyzed (Participants) | 3
percentage of participants | 0.0 [0.0 to 0.0]

2. Primary Outcome: PSA Response 1, Defined as >= 90% PSA Decline From Baseline
Description: The percentage of participants with a >= 90% PSA decline from baseline will be reported with 95% confidence interval using exact method. 'PSA response' is based on Prostate Cancer Working Group 2's (PCWG2) recommendations, which do not offer a specific definition as no single degree of decline has been established.
Time Frame: Baseline to time of >= 90% PSA decline, assessed up to 68 weeks
Population: Phase I and Phase II participants with mCRPC who received at least one cycle of study drugs. For efficacy outcomes, Phase I and II arms were combined as participants in each arm received identical treatments of 25 mg/m2 cabazitaxel q3 weeks plus enzalutamide 160 mg QD. Per protocol, dose limiting toxicities (DLTs) identified during Phase I informed the dose of cabazitaxel in Phase II. No DLTs were identified during Phase I, and the study proceeded to Phase II at the identical dose.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Phase I and Phase II - Treatment (Cabazitaxel, Enzalutamide): Patients receive 25 mg/m2 cabazitaxel IV over 1 hour on day 1 and enzalutamide PO QD on days 1-21 (days 2-21 of cycle 1). Patients also receive prednisone PO BID as standard of care with cabazitaxel. Cycles repeat every 21 days for 6-10 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue enzalutamide PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
  Cabazitaxel: Given IV
  Enzalutamide: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Prednisone: Given PO
Arm/Group | Phase I and Phase II - Treatment (Cabazitaxel, Enzalutamide)
Number analyzed (Participants) | 36
percentage of subjects | 55.6 [38.1 to 72.1]
Statistical Analysis 1: Comparison: Phase I and Phase II - Treatment (Cabazitaxel, Enzalutamide); One-sample binomial test with null hypothesis that the percentage of participants with PSA response 1 is equal to 25%; Test type: Other; p < 0.01, two-sided exact binomial test

3. Secondary Outcome: Incidence of Adverse Events Graded by National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0
Description: Descriptive statistical analysis will be conducted. The proportion estimate will be reported with 95% confidence interval using exact method.
Time Frame: Up to 28 days after the last dose of study medication
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: Descriptive statistical analysis will be conducted. The median overall survival will be estimated with 95% confidence interval (if available). Kaplan-Meier plot will be used to graphically illustrate the overall survival distribution.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Pharmacokinetic Parameters of Cabazitaxel: Max Plasma Concentration (Cmax)
Description: Mean plasma concentration (Cmax) will be plotted over time for cabazitaxel (day 1, cycle 1) and cabazitaxel co-administered with enzalutamide (day 1, cycle 2). Noncompartmental pharmacokinetic analysis will be performed on individual concentration-time data to calculate maximum concentration from 0 hours to last measurable concentration and to infinity, and half-life, for cabazitaxel administered alone or coadministered with enzalutamide.
Time Frame: Day 1 at 0.5, 1, 1.5, 2, 4, 8, and 24 hours after the start of cabazitaxel infusion of cycles 1 and 2 (each cycle is 21 days)
Reporting Status: Not Posted

6. Secondary Outcome: Pharmacokinetic Parameters of Cabazitaxel: Mean Area Under the Curve (AUC)
Description: Mean area under the curve (AUC) will be plotted over time for cabazitaxel (day 1, cycle 1) and cabazitaxel co-administered with enzalutamide (day1, cycle 2). Noncompartmental pharmacokinetic analysis will be performed on individual concentration-time data to calculate AUC from 0 hours to last measurable concentration for cabazitaxel administered alone or coadministered with enzalutamide.
Time Frame: as for outcome 5
Reporting Status: Not Posted

7. Secondary Outcome: Pharmacokinetic Parameters of Cabazitaxel: Mean Cabazitaxel Half-Life
Description: Mean cabazitaxel half-life will be plotted over time for cabazitaxel (day 1, cycle 1) and cabazitaxel co-administered with enzalutamide (day1, cycle 2). Noncompartmental pharmacokinetic analysis will be performed on individual concentration-time data to calculate half-life from 0 hours to last measurable concentration for cabazitaxel administered alone or coadministered with enzalutamide.
Time Frame: as for outcome 5
Reporting Status: Not Posted

8. Secondary Outcome: PSA Response 2, Defined as >= 50% PSA Decline From Baseline
Description: The percentage of participants with a >= 50% PSA decline from baseline will be reported with 95% confidence interval using exact method. 'PSA response' is based on Prostate Cancer Working Group 2's (PCWG2) recommendations, which do not offer a specific definition as no single degree of decline has been established.
Time Frame: Baseline to time of >= 50% PSA decline, assessed up to 68 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Phase I and Phase II - Treatment (Cabazitaxel, Enzalutamide)
Number analyzed (Participants) | 36
percentage of subjects | 77.8 [60.8 to 89.9]

9. Secondary Outcome: PSA Response 3, Defined as >= 30% PSA Decline From Baseline
Description: The percentage of participants with a >= 30% PSA decline from baseline will be reported with 95% confidence interval using exact method. 'PSA response' is based on Prostate Cancer Working Group 2's (PCWG2) recommendations, which do not offer a specific definition as no single degree of decline has been established.
Time Frame: Baseline to time of >= 30% PSA decline, assessed up to 68 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Phase I and Phase II - Treatment (Cabazitaxel, Enzalutamide)
Number analyzed (Participants) | 36
percentage of subjects | 80.6 [64.0 to 91.8]

ADVERSE EVENTS:
Time Frame: Adverse events are recorded from the start of treatment administration to 30 days post treatment or resolution of the event, an average of 20 months.
Description: All adverse events, regardless of causality or relationship to study treatments or procedures, are reported.
Arm/Group | Phase I - Treatment (Cabazitaxel, Enzalutamide) | Phase II - Treatment (Cabazitaxel, Enzalutamide)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/3 | 10/33
Other Adverse Events (participants affected / at risk) | 3/3 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Treatment (Cabazitaxel, Enzalutamide) (N=3) | Phase II - Treatment (Cabazitaxel, Enzalutamide) (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 2
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, influenza (Infections and infestations) | 1 | 0
Myelitis (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (General disorders) | 0 | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 | 1
hematuria (Renal and urinary disorders) | 0 | 1
Infections and infestations - Other, Cellulitis (Infections and infestations) | 0 | 1
Surgical and medical procedures- other: Lung Biopsy (Surgical and medical procedures) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Treatment (Cabazitaxel, Enzalutamide) (N=3) | Phase II - Treatment (Cabazitaxel, Enzalutamide) (N=33)
Dysgeusia (Nervous system disorders) | 2 | 8
Fatigue (General disorders) | 3 | 21
Nausea (Gastrointestinal disorders) | 2 | 18
Weight loss (Investigations) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Anemia (Blood and lymphatic system disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 6
Anxiety (Psychiatric disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Cognitive disturbance (Nervous system disorders) | 1 | 4
constipation (Gastrointestinal disorders) | 1 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Creatinine increased (Investigations) | 0 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 18
Dizziness (Nervous system disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Edema limbs (General disorders) | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
fall (Injury, poisoning and procedural complications) | 0 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
fever (General disorders) | 1 | 4
Gait disturbance (General disorders) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Headache (Nervous system disorders) | 0 | 3
Hematuria (Renal and urinary disorders) | 0 | 6
Hot flashes (Vascular disorders) | 0 | 4
Hypertension (Vascular disorders) | 2 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 2
non-cardiac chest pain (General disorders) | 0 | 4
Pain (General disorders) | 0 | 10
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 12
Platelet count decreased (Investigations) | 0 | 3
Restlessness (Psychiatric disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 5
Urinary tract infection (Infections and infestations) | 1 | 3
Urinary tract pain (Renal and urinary disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 5
Watering eyes (Eye disorders) | 0 | 5
Weight gain (Investigations) | 0 | 3
White blood cell decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 2
Lymphocyte count decreased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
blurred vision (Eye disorders) | 0 | 2
bone pain (Musculoskeletal and connective tissue disorders) | 1 | 4
chills (General disorders) | 0 | 2
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 1 | 1
pelvic pain (Reproductive system and breast disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 2
Urinary urgency (Renal and urinary disorders) | 0 | 2
vertigo (Ear and labyrinth disorders) | 0 | 3
ataxia (Nervous system disorders) | 1 | 0
cataract (Eye disorders) | 1 | 0
Gastrointestinal disorders - Other, Diverticulitis (Gastrointestinal disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Renal and urinary disorders - Other, nocturia (Renal and urinary disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT02522715/Prot_SAP_000.pdf